CLINICAL TRIAL: NCT04769648
Title: A Phase II/III Trial of Safety and Efficacy of Pro-ocular™ 1% in Daily Scleral Lens Wearing Patients With Ocular Graft-versus-Host Disease
Brief Title: Safety and Efficacy of Pro-ocular™ 1% in Daily Scleral Lens Wearing Patients With Ocular Graft-versus-Host Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glia, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: oGvHD-2-SC
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ocular Graft-versus-host Disease
Keywords: scleral lens; scleral lenses; scleral lens wear

STUDY DESIGN:
Intervention Model Description: 12 weeks randomized 1:1 active to placebo. At 12 weeks, placebo group crosses over to active drug. At week 24, all subjects can opt in to an open-label phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects randomized for week 0 - week 12; subjects, investigators and study staff will be masked through week 24.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo
- Pro-ocular™ Topical Gel 1% (Experimental)
  Interventions: Drug: Pro-ocular™ Topical Gel 1%

INTERVENTIONS:
Drug: Pro-ocular™ Topical Gel 1% — Pro-ocular™ is a topical gel applied dermally to forehead twice-daily
  Arms: Pro-ocular™ Topical Gel 1%
Drug: Placebo — Placebo is a vehicle topical gel without active ingredient applied dermally to forehead twice-daily
  Arms: Vehicle

SUMMARY:
This clinical study seeks to evaluate the safety and efficacy of Pro-ocular™1% topical gel in patients with ocular Graft-versus-Host Disease who wear scleral lenses daily. This vehicle-controlled trial will evaluate the investigational drug's effect on signs and symptoms of ocular Graft-versus-Host Disease and on the hours of daily comfortable and serviceable scleral lens wear.

DETAILED DESCRIPTION:
This Phase 2/3 placebo-controlled clinical study of Safety and Efficacy of Pro-ocular™ 1% in Daily Scleral Lens Wearing Patients with Ocular Graft-versus-Host Disease (oGvHD) will evaluate the the investigational drug's effect on signs and symptoms of oGvHD and subject-reported hours of duration of comfortable and serviceable scleral lens wear time.

The study will enroll 38 subjects. In the first 12 weeks, subjects will be randomized 1:1 active to placebo. At week 12, placebo subjects will cross-over to active drug treatment. At week 24, all subjects can opt into an open label phase.

In clinic visits will occur at weeks 0, 12 and 24 with remote telephone assessments at weeks 6 and 18. For subjects who opt into the open-label phase, in-clinic visits will occur at weeks 36 and 52.

Safety monitoring for adverse events will be performed at all onsite and remote visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race, at least 18 years of age at Visit 1.
2. Has had the diagnosis of ocular GvHD (oGvHD) for at least 3 months prior to Visit 1.
3. Use of scleral lenses daily in both eyes for at least two months prior to Visit 1 for treatment of oGvHD with planned continuation for use of the same scleral lenses throughout this study.
4. Excluding final scleral lens removal of the day, after successful daily insertion, patient feels need to remove or does remove one or both scleral lenses at least once per day due to physical discomfort or visual acuity issues (lenses have debris or deposit build up or vision is foggy, cloudy or blurry).
5. Has staining score in central corneal region of ≥ 2 out of 10 in either eye at Visit 1.
6. Has Modified SANDE Frequency score of ≥ 35 out of 100 in either eye for both Modified SANDE daytime questionnaire with lenses and Modified SANDE nighttime questionnaire without lenses.
7. Has provided verbal and written informed consent.
8. Be able and willing to follow oral and written instructions provided in English, with or without assistance and participate in all assessments and visits.
9. Has access to telephone necessary for evaluations.
10. Had an ophthalmological exam within past year prior to Visit 1.

Exclusion Criteria:

1. Has tested positive from COVID-19 within twenty-eight days prior to Screening.
2. Active trigeminal neuritis, trigeminal neuralgia, ocular herpes zoster, facial herpes zoster, ocular herpes simplex, or neurotrophic keratitis at Visit 1.
3. History of ocular herpes zoster, facial herpes zoster, ocular herpes simplex, or neurotrophic keratitis within the last 5 years that is not being medically managed including oral antivirals. Patients with a history of herpes simplex virus must be receiving appropriate antiviral therapy.
4. History of breast cancer in patient or immediate biological family (parents, siblings and children).
5. Eyelid surgery or ocular surgery within the last 12 weeks prior to screening that in the judgment of the clinical investigator will interfere with study assessments.
6. Comorbidity with other severe, acute or chronic systemic or ocular condition that in the judgment of the investigator will interfere with study assessments, study participant safety, or study compliance such as active COVID-19 infection.
7. Significant change (e.g. discontinuation) in oral corticosteroid dose or corticosteroid-containing eye drops or gels, cyclosporine ophthalmic emulsion or lifitegrast ophthalmic solution within 7 days prior to screening.
8. Wears any type of lenses overnight (e.g. scleral lenses, bandage contact lenses).
9. Women of childbearing potential who are pregnant, nursing an infant, planning a pregnancy, not receiving an adequate method of birth control, or have a positive urine pregnancy test at Screening. Women of childbearing potential must be willing to use contraception throughout this study.
10. Has a known adverse reaction and/or sensitivity to the study drug.
11. Prior or current use of Pro-ocular™.
12. Unwilling to cease the use of sunscreen on the forehead or eye area.
13. Currently using more than one preserved topical medication for glaucoma.
14. Currently enrolled in an investigational drug or device study exclusively for ocular GvHD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Symptom Assessment in Dry Eye Questionnaire, Global Score for nighttime without scleral lenses. | 12 weeks
  0-100 visual analog scale, lower score is a better outcome than a higher score

SECONDARY OUTCOMES:
Change in Central Corneal Staining | 12 weeks
  0-10 scale, lower score is a better outcome than a higher score
Change in Blurred or Cloudy Vision in Glia Ocular Surface Disease Symptoms Questionnaire. | 12 weeks
  0-10 scale, lower score is a better outcome than a higher score

OTHER OUTCOMES:
Change in Corneal fluorescein staining using modified NEI scoring. | 12 weeks
  0-10 scale, lower score is a better outcome than a higher score
Change in Conjunctival lissamine staining using NEI scoring. | 12 weeks
  0-10 scale, lower score is a better outcome than a higher score
Change in Eyelid evaluation using Efron scale with 0.5 steps (with and without scleral lenses). | 12 weeks
  0-4 scale with 0.5 steps, lower score is a better outcome than a higher score
Change in Conjunctival redness using Efron scale with 0.5 steps (with and without scleral lenses). | 12 weeks
  0-4 scale with 0.5 steps, lower score is a better outcome than a higher score
Change in Tear break-up time using fluorescein and slit lamp. | 12 weeks
  0-10 scale, higher score is a better outcome than a lower score
Change in Eye redness using redness scan by keratograph. | 12 weeks
Change in Modified Glia Ocular Surface Disease Symptoms Questionnaire using VAS. | 6 weeks, 12 weeks
  patient-reported ocular discomfort, dryness, conjunctival redness, photophobia, blurred or cloudy vision, difficulty blinking and level of sleep disturbance; 0-10 visual analog scale, lower score is a better outcome than a higher score
Change in Scleral Lens Wear Glia Questionnaire | 6 weeks, 12 weeks
  total hours daily scleral lens wear, daily hours of comfort wear, daily hours of serviceable wear, number of instances of lens removal for cleaning and re-insertion.
Change in Modified Symptom Assessment in Dry Eye Questionnaire in daytime with scleral lenses and at nighttime without scleral lenses. | 6 weeks, 12 weeks
  0-100 scale, lower score is a better outcome than a higher score

CONTACTS AND LOCATIONS:
Locations (1):
- BostonSight, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No